CLINICAL TRIAL: NCT02744144
Title: Wound Bacterial Microbiota and Their Antibiotic Resistance: a Prospective Cohort Study of Hospitalized Patients Originating From the Syrian Armed Conflict
Brief Title: Wound Bacterial Microbiota and Their Antibiotic Resistance
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Principal Investigator, Jonas Malmstedt, co-pi, Karolinska Institutet
Other Study IDs: KISOS002
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Wounds and Injuries; War-Related Injuries; Wound Infection; Wounds, Penetrating; Wounds, Gunshot; Arm Injuries; Leg Injuries; Soft Tissue Injuries
MeSH Terms: conditions — Wounds and Injuries; War-Related Injuries; Wound Infection; Wounds, Penetrating; Wounds, Gunshot; Arm Injuries; Leg Injuries; Soft Tissue Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-infection: Patients without clinical infection or positive wound culture
- Infection: Patients with clinical infection and positive wound culture

SUMMARY:
The purpose of the study is to explore the microbiology in war-associated wounds of hospitalized patients from the Syrian armed conflict. Cultures collected from acute wounds with clinical signs of infection will be analyzed.

DETAILED DESCRIPTION:
War-associated injuries often result in soft tissue and bone being contaminated with foreign material, leading to infection (Fares et al. 2013; Covey, Lurate, and Hatton 2000). Wound infections remain the greatest risk to life and restoration of function in war-wounded that survive the first few hours (Tong 1972; Murray 2008).

The Syrian armed conflict broke out in 2011 and quickly deteriorated. Médecins Sans Frontières/Doctors Without Borders (MSF) runs an emergency trauma project in the Ministry of Health hospital in Ar Ramtha, Jordan, less than five kilometers from the Syrian border. At this facility patients from the Syrian armed conflict receive treatment for blast- and gunshot-injuries. Wounds are treated according to the International Committee of the Red Cross war surgery protocol (Giannou and Baldan 2010). Wound management and healing has been difficult and time consuming, often complicated by infections and antibiotic resistance.

Recommendations for treatment of war-associated infections are generally not supported by cohort studies (Murray et al. 2008). High rates of war wound infections caused by antimicrobial drug resistant organisms have been shown in the Middle East but reports generally only include combatants. Due to the use of body armor and forward medical therapy this data may not be applicable to a civilian setting. Furthermore, available studies are either performed on old wounds (Teicher et al. 2014) or on all available culture samples, disregarding infection signs (Sutter et al. 2011; Dau, Tloba, and Daw 2013). Without clinical signs of infection, routine collection of peri-debridement culture samples is inappropriate in war-associated injuries (Murray et al. 2008). The differentiation between contamination and infecting organisms is crucial in order to avoid unnecessary medication, especially limit the use of broad-spectrum antibiotics as overuse may lead to development of multi-drug resistant organisms (Eardley et al. 2011). Cultures collected from acute wounds with clinical signs of infection will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients that receive surgical treatment for war-associated injuries, irrespective of injury location, injury mechanism, time from injury and prior treatment
* Patients that receive treatment during the study period and are later re-admitted will only be counted as one patient

Exclusion Criteria:

* Patients that are only re-admitted during the study period, i.e. patients that received primary treatment by MSF before study initiation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients originating from the Syrian armed conflict who receive treatment for blast- and gunshot-injuries.
Sampling Method: Non-Probability Sample
Enrollment: 457 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that develops infections after receiving surgical treatment | 30 days

SECONDARY OUTCOMES:
Frequency of different bacterial microbiota in wounds with clinical signs of infection | 30 days
  For wounds with clinical signs of infection the bacterial microbiota will be characterized.
Frequency of microbiota with antibiotic resistance in wounds with clinical signs of infection | 30 days
  For wounds with clinical signs of infection the the antibiotic resistance patterns of the bacterial microbiota will be characterized.
Length of stay | 30 days
  Length of hospital stay
Surgery | 30 days
  Number and type of surgeries
Death | 30 days
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Malmstedt, MD, PhD, Study Director — Karolinska Institutet
Locations (1):
- Ministry of Health hospital, Ar Ramtha, Irbid Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fares Y, El-Zaatari M, Fares J, Bedrosian N, Yared N. Trauma-related infections due to cluster munitions. J Infect Public Health. 2013 Dec;6(6):482-6. doi: 10.1016/j.jiph.2013.05.006. Epub 2013 Jul 31. PMID 23999350
- [Background] Covey DC, Lurate RB, Hatton CT. Field hospital treatment of blast wounds of the musculoskeletal system during the Yugoslav civil war. J Orthop Trauma. 2000 May;14(4):278-86; discussion 277. doi: 10.1097/00005131-200005000-00010. PMID 10898201
- [Background] Tong MJ. Septic complications of war wounds. JAMA. 1972 Feb 21;219(8):1044-7. No abstract available. PMID 4621762
- [Background] Murray CK. Infectious disease complications of combat-related injuries. Crit Care Med. 2008 Jul;36(7 Suppl):S358-64. doi: 10.1097/CCM.0b013e31817e2ffc. PMID 18594263
- [Background] Giannou C, Baldan M. War Surgery: Working With Limited Resources in Armed Conflict and Other Situations of Violence. ICRC; 2010.
- [Background] Murray CK, Hsu JR, Solomkin JS, Keeling JJ, Andersen RC, Ficke JR, Calhoun JH. Prevention and management of infections associated with combat-related extremity injuries. J Trauma. 2008 Mar;64(3 Suppl):S239-51. doi: 10.1097/TA.0b013e318163cd14. PMID 18316968
- [Background] Teicher CL, Ronat JB, Fakhri RM, Basel M, Labar AS, Herard P, Murphy RA. Antimicrobial drug-resistant bacteria isolated from Syrian war-injured patients, August 2011-March 2013. Emerg Infect Dis. 2014 Nov;20(11):1949-51. doi: 10.3201/eid2011.140835. No abstract available. PMID 25340505
- [Background] Sutter DE, Bradshaw LU, Simkins LH, Summers AM, Atha M, Elwood RL, Robertson JL, Murray CK, Wortmann GW, Hospenthal DR. High incidence of multidrug-resistant gram-negative bacteria recovered from Afghan patients at a deployed US military hospital. Infect Control Hosp Epidemiol. 2011 Sep;32(9):854-60. doi: 10.1086/661284. PMID 21828965
- [Background] Dau AA, Tloba S, Daw MA. Characterization of wound infections among patients injured during the 2011 Libyan conflict. East Mediterr Health J. 2013 Apr;19(4):356-61. PMID 23882961
- [Background] Eardley WG, Brown KV, Bonner TJ, Green AD, Clasper JC. Infection in conflict wounded. Philos Trans R Soc Lond B Biol Sci. 2011 Jan 27;366(1562):204-18. doi: 10.1098/rstb.2010.0225. PMID 21149356
- [Derived] Alga A, Wong S, Shoaib M, Lundgren K, Giske CG, von Schreeb J, Malmstedt J. Infection with high proportion of multidrug-resistant bacteria in conflict-related injuries is associated with poor outcomes and excess resource consumption: a cohort study of Syrian patients treated in Jordan. BMC Infect Dis. 2018 May 22;18(1):233. doi: 10.1186/s12879-018-3149-y. PMID 29788910